CLINICAL TRIAL: NCT03198338
Title: Ultrasound Guided Transversus Abdominis Plane(TAP) Block in Intensive Care Unit(ICU) for Postoperative Analgesia After Open Colon Resection: a Double Blind Randomized Controlled Trial
Brief Title: Ultrasound Guided Transversus Abdominis Plane(TAP) Block in Intensive Care Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Tak Kyu Oh, Clinical Professor of Anesthesiology and Pain department, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B1706-401-001
Record Dates: First submitted 2017-06-20; First posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Colon Neoplasm; Rectum Neoplasm; Perforated Colon; Perforated Bowel
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Intestinal Perforation | interventions — Bupivacaine; Saline Solution; Ultrasonography

STUDY DESIGN:
Intervention Model Description: Randomized Double Blind study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Drugs that are not directly involved in the study are delivered to the practitioner without specific labeling of the drug to be used in the block. The practitioner, the patient, and the observer all undergo TAP block without knowing which group the patient belongs to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP group (Experimental): Drug: 0.25% Bupivacaine, 0.5mL/kg
  Interventions: Drug: 0.25% Bupivacaine, 0.5mL/kg; Device: Ultrasound
- Placebo group (Sham Comparator): Drug: 0.9% Normal Saline, 0.5mL/kg
  Interventions: Drug: Normal Saline; Device: Ultrasound

INTERVENTIONS:
Drug: 0.25% Bupivacaine, 0.5mL/kg — Ultrasound guided TAP block using 0.25% Bupivacaine, 0.5ml/kg
  Arms: TAP group
Drug: Normal Saline — 0.9% Normal Saline
  Arms: Placebo group
Device: Ultrasound — Ultrasound guided TAP block

SUMMARY:
The Transversus Abdominis Block (TAP) block is known to be an effective means of reducing patient pain after abdominal surgery. In the meantime, the general TAP block has been studied in patients who were in the recovery room and the ward after surgery. The purpose of this study was to determine the effect of pain reduction and opioid saving effects in patients with TAP block in ICU settings.

DETAILED DESCRIPTION:
This study is a prospective study in a single institute of Seoul National University Bundang Hospital and is assigned to the test group and the control group by random assignment. In both groups, PCA (Patient Controlled Analgesia) was used as a post-operative pain control modality. In the Intervention group, a 0.25% Bupivacaine was used for transverse nerve block , and normal saline was used for placebo(control) group

The TAP block will be performed within 1 hour after entering the intensive care unit (ICU) in double blinded state

ELIGIBILITY:
Inclusion Criteria:

* Adults over 20 years of age
* Patients who entered the intensive care unit for monitoring and recovery after colonic resection through laparotomy
* Patients who voluntarily sign a written informed consent and know they have the right to withdraw their consent at any time.

Exclusion Criteria:

* Patients who are unconscious and require sedation below the Richmond Agitation Sedation Scale (-2) Patients who need continuous renal replacement therapy, cardiopulmonary bypass Patients with a history of allergic reactions to local anesthetics Patients resistant to narcotic analgesics (users of existing long-term narcotic analgesics) Patients who can not use self-analgesic treatment Patients who underwent surgery for organs other than abdomen and pelvis Patients with severe blood clotting disorders with a Prothrombin Time International normalized ratio of 2.0 or greater and Platelet less than 50,000

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
opioid consumption up to 24 hours | 24hour after TAP block
  The total amount of IV Fentanyl (10mcg/cc) used by the patients for 24 hours. Patient Controlled Analgesia will be used.

SECONDARY OUTCOMES:
resting pain score | 2hour, 6hour, 12hour, 24hour after TAP block
  resting Numeric Rating Scale, 0-10, 0= no pain, 10= most severe pain
Nausea score | 2hour, 6hour, 12hour, 24hour after TAP block
  Nausea score, 0=none, 1=nausea symptom, 2- nausea requiring treatment, 3=vomiting
sedation score | 2hour, 6hour, 12hour, 24hour after TAP block
  0- awake, 1- mild sedation, easy to rouse, 1s= asleep, easy to rouse, 2-moderate sedation, unable to remain awake, 3- difficult to rouse

CONTACTS AND LOCATIONS:
Overall Officials: In Ae Song, M.D. Ph.D., Principal Investigator — Department of Anesthesiology and Pain Medicine, Seoul National University Bundang Hospital
Locations (1):
- Department of Anesthesiology and Pain department, Seongnam-si, Gyeong Gi Do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
It can be shared after request to principal investigator (T.K Oh or I.A Song)

REFERENCES:
- [Background] Niraj G, Kelkar A, Fox AJ. Application of the transversus abdominis plane block in the intensive care unit. Anaesth Intensive Care. 2009 Jul;37(4):650-2. doi: 10.1177/0310057X0903700420. PMID 19681428